CLINICAL TRIAL: NCT01045551
Title: An Open Label, Pilot Study to Determine the Efficacy of Apremilast in the Treatment of Rosacea in Patients With Both Erythematotelangiectatic Rosacea and Papulopustular Rosacea
Brief Title: Open Label Pilot Study of Apremilast in Treatment of Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Julian M. Mackay-Wiggan (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Julian M. Mackay-Wiggan, Assistant Clinical Professor of Dermatology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAE1745; AP-ROS-PI 0033 (Other: Celgene)
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: Erythematotelangiectatic Rosacea; Papulopustular Rosacea
Keywords: Inflammatory rosacea; Papules and pustules; Moderate to severe erythema; Telangiectasia
MeSH Terms: conditions — Rosacea; Telangiectasis | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apremilast 20 mg (twice per day) (Experimental): All subjects will receive Apremilast 20mg taken orally twice per day.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — 20mg taken orally twice per day for 12 weeks

SUMMARY:
Rosacea is a chronic skin disorder with the signs and symptoms of facial flushing, persistent redness, small visible spider-like veins, papules (inflamed red bumps under the skin) and pustules. Rosacea is also a a recurring skin disorder. In addition to causing uncomfortable and embarrassing physical symptoms such as flushing, burning, and itching, rosacea can also contribute to lower self-esteem, which can have a significant psychosocial impact on quality of life. Rosacea flares can be triggered by every day factors such as sun exposure, heat, hot or caffeinated drinks, alcoholic beverages, spices and stress.

Many of the currently available treatments for rosacea are only partially effective and some patients do not respond to them, or are unable to tolerate the side effects.

This is a single-center, open label trial of Apremilast in ten (10) subjects with moderate to severe inflammatory rosacea who will be treated with Apremilast 20 mg twice per day for 12 weeks. Following the screening period and baseline visit, study subjects will return at weeks 1, 2, 4, 6, 8, 10 and 12. There is a follow up study visit at week 16.

Recent research has shown an increase of specific proinflammatory cytokines in the biopsies of inflammatory lesions from rosacea and acne patients. The cytokines then trigger a chain of chemical responses in the body that likely result in the development of the papules an pustules that are seen in rosacea and acne patients. Apremilast is an oral agent that modulates multiple anti-inflammatory pathways and has pharmacodynamic properties with potential therapeutic benefit for treating inflammatory autoimmune disorders.

The investigators therefore propose a pilot study to evaluate the potential for Apremilast to improve the signs and symptoms of moderate to severe inflammatory rosacea.

DETAILED DESCRIPTION:
This is a single-center, open label pilot study of Apremilast in ten subjects with both erythematotelangiectatic rosacea and papulopustular rosacea in which subjects will be treated with Apremilast 20mg twice per day for 12 weeks. There is a total of 10 visits over a period of 16 weeks.

Adult male and female subjects 18 years of age or older will participate in the study after the objectives, methods, and potential hazards of the study have been fully explained, and after they have signed the informed consent form. Subjects must have a diagnosis or findings consistent with erythematotelangiectatic and papulopustular rosacea. Subjects must have at least 10 papulopustular lesions with underlying erythema/telangiectasias visible to the unassisted naked eye.

Subjects will take Apremilast capsules 20mg twice per day for 12 weeks. If at anytime during the study a subject encounters overt study medication related adverse effects, dose reduction will be allowed following discussions between the subject and the investigator. Dose reductions to 20mg once per day will be allowed for subjects who experience intolerable adverse effects from the study medication. If the subject cannot tolerate 20mg per day, he/she will be terminated from the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be a healthy, post-pubescent male or female 18 years of age or older with moderate to severe erythematotelangiectatic and papulopustular rosacea, defined as 10 to 40 papules and pustules
* Must have presence of moderate to severe erythema
* Must have presence of telangiectasia
* Must have a diagnosis or findings consistent with a diagnosis of erythematotelangiectatic rosacea and papulopustular rosacea
* Must understand and voluntarily sign an informed consent form
* Must be ale to adhere to the study visit schedule and other protocol requirements
* Must be able to restrict diet in order to avoid foods/drinks that are known triggers that would exacerbate the signs/symptoms of rosacea
* Must have within normal range for routine blood laboratory tests
* Females of childbearing potential must have a negative urine pregnancy test at screening and if sexually active must agree to use two(2) forms of contraception (adequate forms of contraception are outlined in the protocol)
* Females of childbearing potential must agree to serum pregnancy tests every 4 weeks while on study medication
* Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in sexual activity with females of childbearing potential while on study medication and for 84 days after taking the last dose of study medication

Exclusion Criteria:

* Inability to provide voluntary consent
* Diagnosis of acne vulgaris or perioral dermatitis
* Use of topical acne or rosacea treatments within 4 weeks of baseline
* Use of systemic retinoids within 90 days of baseline
* Known or suspected excessive alcohol intake (which in the opinion of the investigator will exacerbate the signs and symptoms of rosacea)
* Use of any investigational medication within 4 weeks prior to start of study drug or 5 pharmacokinetic/pharmacodynamic half-lives (whichever is longer)
* A known sensitivity to tetracyclines
* Currently taking clinically significant concomitant drug therapy
* Use of any acne or rosacea treatment during the course of the study or within four weeks of starting the study medication, including azelaic acid, topical or systemic retinoids, sulfa drugs, erythromycin, cephalosporins, quinolones, tetracycline, benzoyl peroxide products, as well as pulse dye laser, intense pulsed light and photodynamic therapy
* Current use and inability to discontinue use of PDE 4 inhibitors, theophylline, systemic steroids (oral or inhaled), penicillin antibiotics, niacin greater than 500 mg/day, chronic use of NSAIDS, or use of any medication that in the opinion of the investigator affects the severity of rosacea
* Long-term use (greater than 14 days) of topical or systemic anti-inflammatories in the 4 weeks prior to baseline and during the study. Chronic use of aspirin at sub-analgesic doses (less than 325 mg once daily) is acceptable for patients requiring platelet aggregation inhibition
* Use of topical or systemic corticosteroids 4 weeks prior to baseline and during the study
* Patients with ocular rosacea and/or blepharitis/meibomianitis who required treatment by an ophthalmologist
* Patients who had surgeries that bypassed or excluded the duodenum
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Pregnant or breastfeeding women, or women of childbearing potential who are not using an adequate form of birth control as described in the inclusion criteria
* Initiation of a hormonal method of birth contraception within 4 months of baseline, discontinuation during the course of the study, or change in the product within 4 months of baseline during the study
* Subject is a woman who is perimenopausal whos symptoms cause flushing that may affect the rosacea
* Systemic fungal infection
* History of active mycobacterial infection with any species within 3 years prior to screening, subjects with mycobacterium tuberculosis infection more than 3 years prior to screening are allowed if successful treatment was completed at least 3 years prior to randomization and is documented and available for verification
* Latent mycobacterium tuberculosis infection as indicated by a positive purified protein derivative (PPD) skin test. Subjects with a positive PPD skin test and documented completion of treatment for latent TB are eligible. Subjects with a positive PPD skin test and not treated or no documentation of completion of treatment are ineligible
* History of incompletely treated mycobacterium tuberculosis infection as indicated by: a)subject's medical records documenting incomplete treatment for mycobacterium tuberculosis b)subject's self reported history of incomplete treatment for mycobacterium tuberculosis
* History of recurrent bacterial infection (at least 3 major infections resulting in hospitalization and/or requiring intravenous antibiotic treatment within the past 2 years)
* Clinically significant abnormality on the chest x-ray at screening, chest x-rays performed within 3 months prior to start of study drug are acceptable
* Any clinically significant abnormality on 12-lead electrocardiogram at screening
* History of congenital or acquired immunodeficiency (common variable immunodeficiency (CVID) Hepatitis B surface antigen positive or Hepatitis B core antibody positive at screening
* History of human immunodeficiency virus (HIV) infection
* Antibodies to hepatitis C at screening
* Malignancy or history of malignancy (except for treated/cured basal cell skin carcinoma) greater than 3 years prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Mackay-Wiggan, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 patients recruited
Period: Overall Study
Arm/Group | Apremilast 20 mg (Twice Per Day)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Apremilast 20 mg (Twice Per Day)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Gender [Count of Participants; unit: Participants]
  Female | 7
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Number of Papulopustular Lesions at Week 12
Description: Papule and pustule count consisted of direct measurement of the number of papules/pustules on the face. Papule and pustule count, compared between baseline and end of treatment Week 12 was calculated
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: papule count
Groups:
- Open Label Apremilast 20 mg (Twice Per Day): This is an open label study, therefore all subjects will receive Apremilast 20mg taken orally twice per day.
  Apremilast: 20mg taken orally twice per day for 12 weeks
Arm/Group | Open Label Apremilast 20 mg (Twice Per Day)
Number analyzed (Participants) | 10
papule count | -0.2 (25.77165)
Statistical Analysis 1: Comparison: Open Label Apremilast 20 mg (Twice Per Day); Test type: Superiority or Other; p = 0.98, t-test, 2 sided — The a priori threshold for statistical significance was P<0.05; Mean Difference (Final Values) = -0.2

2. Secondary Outcome: Change in Physician 7 Point Global Assessment From Baseline to Week 12
Description: The Physician Global 7-point Assessment. Scale range: 0-7. 0 = clear, 1 = minimal, 2 = mild, 3 = mild to moderate, 4= moderate, 5= moderate to severe, 6 = severe. 0 is a better outcome, 6 is a worse outcome. No subscales were used.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 20 mg (Twice Per Day)
Number analyzed (Participants) | 10
units on a scale | -0.90000 (0.99443)
Statistical Analysis 1: Comparison: Apremilast 20 mg (Twice Per Day); Test type: Superiority or Other; Mean Difference (Net) = 0.09, Standard Deviation 0.9024

3. Secondary Outcome: Change From Baseline in Erythema Rating Visit 8 (Week 12)
Description: The change in the Physician Overall Erythema Severity. Scale range 0 - 3. 0 = none/absent, 1 = mild, 2 = moderate, 3 = severe. 0 is considered a better outcome, 3 is considered a worse outcome.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast 20 mg (Twice Per Day)
Number analyzed (Participants) | 10
units on a scale | -0.7000 (0.48305)

4. Secondary Outcome: Change From Baseline in Telangiectasia Count at Visit 8 (Week 12)
Description: physician count of telangiectasias on the face at visit 1 (baseline) compared to at visit 8 (week 12)
Time Frame: Baseline, Week 12
Measure: Mean (Standard Error); unit: telangiectasia count
Arm/Group | Open Label Apremilast 20 mg (Twice Per Day)
Number analyzed (Participants) | 10
telangiectasia count | 0 (0)

5. Secondary Outcome: Change From Visit 8 (Week 12) in Telangiectasia Count at Visit 9 (Week 16)
Time Frame: Week 12, Week 16
Measure: Mean (Standard Error); unit: telangiectasia count
Arm/Group | Open Label Apremilast 20 mg (Twice Per Day)
Number analyzed (Participants) | 10
telangiectasia count | 0.2000 (0.63246)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for approximately 4 years.
Description: Adverse event determination was achieved by regular solicitation subjects at study visits, from investigator assessment, and regular laboratory testing.
  In addition self-reporting by participants was encouraged.
Groups:
- Apremilast 20 mg (Twice Per Day): All subjects will receive Apremilast 20mg taken orally twice per day.
  Apremilast: 20mg taken orally twice per day for 12 weeks
  The most frequently reported adverse event (AE) was infection. One patient (a 74 year old female) experienced 2 urinary tract infections during the course of the study, and another (a 63 year old female) experienced one urinary tract infection. Two patients experienced upper respiratory infections, which have previously been reported in patients taking apremilast. The second most common AE was loose stool, reported by two patients, which resolved quickly and without recurrence. All AE's were reported as mild and no patient withdrew from the study due to AEs. No patient required dosing modification or discontinuation.
Arm/Group | Apremilast 20 mg (Twice Per Day)
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast 20 mg (Twice Per Day) (N=10)
urinary tract infection (Renal and urinary disorders) | 2 (3)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
loose stool (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes